CLINICAL TRIAL: NCT03716219
Title: Exercise Training in Children and Adults: Mechanisms of Allaying Inflammation in Asthma
Brief Title: The Effect of 10-Week Exercise Training on Children With Asthma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Nonapplicable clinical trial
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2012-9253
Record Dates: First submitted 2018-10-03; First posted 2018-10-23 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Asthma in Children
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Subjects (Other): Healthy control group which received the same exercise training intervention as the experimental group
  Interventions: Other: Exercise Training
- Subjects with Asthma (Experimental): Subjects with asthma who received exercise training
  Interventions: Other: Exercise Training

INTERVENTIONS:
Other: Exercise Training — Physical activity in children and adults with asthma.

SUMMARY:
The goal of this research is to determine whether 10-weeks of exercise training can benefit asthmatic children and young adults with a history of exercise-induced bronchoconstriction (EIB). The investigators will also study an exciting newly discovered aspect of gene expression regulation in the white blood cells known as epigenetics: a process that takes place when genomic changes happen as a result of exposure to the environment. This study is based on emerging exciting new data from this and other laboratories demonstrating that (a) white blood cells play an important role in bronchoconstriction in children, (b) gene and cytokine expression in circulating white blood cells are abnormal in asthma and (c) brief exercise may change genomic and inflammatory- profiles of these cells.Physical activity is an essential component of growth and health in children, thus, this research will lead to improved clinical uses of exercise as preventive and adjunctive therapy in the current epidemic of childhood asthma

ELIGIBILITY:
Inclusion Criteria:

* Good health
* Physical activity
* No evidence of disease or disability
* Diagnosed with persistent asthma (asthma subjects)
* BMI<95 percentile

Exclusion Criteria:

* Use of illegal drugs or alcohol
* Very high physical fitness
* Pregnancy
* More than two asthma attack per week (asthma subjects)

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10-10 (Actual); Primary Completion 2013-10-10 (Actual); Study Completion 2013-10-10 (Actual)

PRIMARY OUTCOMES:
Gene and microRNA expression will be compared between healthy and asthmatic subjects | 12 weeks
  Monocyte gene expression profiling before and after acute bout of exercise before and after 10-week exercise intervention is gauged using RNA seq in a group of children with asthma and age and sex match healthy controls

SECONDARY OUTCOMES:
Pro/anti-inflammatory cytokines and markers of oxidative stress will be compared between the groups | 12 weeks
  Absolute values of cytokines, growth hormones, and other biomarkers will be measured by flow cytometry and statistically analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Exercise and Genomics Research Center, University of California, Irvine, Irvine, California, United States

REFERENCES:
- [Background] Drews AC, Pizzichini MM, Pizzichini E, Pereira MU, Pitrez PM, Jones MH, Sly PD, Stein RT. Neutrophilic airway inflammation is a main feature of induced sputum in nonatopic asthmatic children. Allergy. 2009 Nov;64(11):1597-601. doi: 10.1111/j.1398-9995.2009.02057.x. Epub 2009 Apr 14. PMID 19392986
- [Background] Dougherty RH, Fahy JV. Acute exacerbations of asthma: epidemiology, biology and the exacerbation-prone phenotype. Clin Exp Allergy. 2009 Feb;39(2):193-202. doi: 10.1111/j.1365-2222.2008.03157.x. PMID 19187331
- [Background] Baines KJ, Simpson JL, Scott RJ, Gibson PG. Immune responses of airway neutrophils are impaired in asthma. Exp Lung Res. 2009 Sep;35(7):554-69. doi: 10.1080/01902140902777490. PMID 19842845
- [Background] Baines KJ, Simpson JL, Bowden NA, Scott RJ, Gibson PG. Differential gene expression and cytokine production from neutrophils in asthma phenotypes. Eur Respir J. 2010 Mar;35(3):522-31. doi: 10.1183/09031936.00027409. Epub 2009 Sep 24. PMID 19797135
- [Background] Radom-Aizik S, Zaldivar F Jr, Oliver S, Galassetti P, Cooper DM. Evidence for microRNA involvement in exercise-associated neutrophil gene expression changes. J Appl Physiol (1985). 2010 Jul;109(1):252-61. doi: 10.1152/japplphysiol.01291.2009. Epub 2010 Jan 28. PMID 20110541
- [Background] Cooper DM, Radom-Aizik S, Schwindt C, Zaldivar F Jr. Dangerous exercise: lessons learned from dysregulated inflammatory responses to physical activity. J Appl Physiol (1985). 2007 Aug;103(2):700-9. doi: 10.1152/japplphysiol.00225.2007. Epub 2007 May 10. PMID 17495117
- [Background] Petersen AM, Pedersen BK. The role of IL-6 in mediating the anti-inflammatory effects of exercise. J Physiol Pharmacol. 2006 Nov;57 Suppl 10:43-51. PMID 17242490

DOCUMENTS (1):
  • Study Protocol (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/19/NCT03716219/Prot_000.pdf